CLINICAL TRIAL: NCT00485550
Title: A Randomized, Double-Blind Comparison of Atomoxetine Hydrochloride Augmented With Either Extended-Release Methylphenidate Hydrochloride (Concerta-TM) or Placebo in Children With Attention-Deficit/Hyperactivity Disorder (ADHD) Who Have Not Responded to Stimulant Mono Therapy
Brief Title: Comparison of Atomoxetine Plus Either Comparator or Placebo in Children With ADHD Who Haven't Responded to Stimulant Therapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 7065; B4Z-MC-LYBU
Record Dates: First submitted 2007-06-11; First posted 2007-06-13 (Estimated); Last update posted 2007-06-13 (Estimated); Status verified 2007-06

CONDITIONS: Attention Deficit Hyperactivity Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Atomoxetine Hydrochloride; Methylphenidate

INTERVENTIONS:
Drug: Atomoxetine Hydrochloride
Drug: Methylphenidate Hydrochloride
Drug: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of atomoxetine alone versus atomoxetine plus low-dose, sustained-release MPH in children with treatment-resistant ADHD.

ELIGIBILITY:
Inclusion Criteria:

* Patients will be at least 6 years of age and not more than 12 years of age at visit 1
* Patients must meet DSM-IV diagnostic criteria for ADHD
* Patients must be retrospectively identified as stimulant non-responders
* Patients must be of normal intelligence as assessed by the investigator (that is, without a general impairment of intelligence and likely, in the investigator's judgment, to achieve a score of greater than or equal to 70 on an IQ test)
* Patients must be able to swallow capsules

Exclusion Criteria:

* Patients who weigh less than 22 kg or more than 60 kg at study entry
* Patients who have a history of Bipolar I or Bipolar II Disorder, psychosis, or pervasive developmental disorder
* Patients who meet DSM-IV criteria for anxiety disorder or autism
* Patients with a history of any seizure disorder and/or Rolandic seizures (other than febrile seizures) or prior electroencephalogram (ECG) abnormalities in the absence of seizures, or patients who have taken (or are currently taking) anticonvulsants for seizure control
* Patients with a history of severe allergies to more than one class of medication or multiple adverse drug reactions, including hypersensitivity to MPH

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 14 (Actual)
Dates: Start 2004-01; Study Completion 2005-03 (Actual)

PRIMARY OUTCOMES:
Assess the safety of atomoxetine and placebo compared to atomoxetine and methylphenidate in children aged 6 through 12 years with ADHD who have been identified as stimulant non-responders and have been exposed to acute treatment of atomoxetine.

SECONDARY OUTCOMES:
Assess the safety of atomoxetine and placebo as compared to atomoxetine and methylphenidate for the treatment of ADHD in children retrospectively identified as stimulant non-responders as measured by ECGs
Assess the safety of atomoxetine and placebo as compared to atomoxetine and methylphenidate for the treatment of ADHD in children retrospectively identified as stimulant non-responders as measured by clinical laboratory tests
Assess the tolerability of atomoxetine and placebo as compared to atomoxetine and methylphenidate for the treatment of ADHD in children retrospectively identified as stimulant non-responders as measured by spontaneously reported AEs
Compare the efficacy of atomoxetine and placebo as compared to atomoxetine and methylphenidate for the treatment of ADHD in children

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Scottsdale, Arizona, United States

REFERENCES:
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com